CLINICAL TRIAL: NCT05280184
Title: Coin2Dose: Behavioral Economics to Promote Insulin BOLUS Activity and Improve HbA1c in Teens
Acronym: Coin2Dose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Susana Patton, Principal Research Scientist, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1770218
Record Dates: First submitted 2022-02-15; First posted 2022-03-15 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coin2Dose (Experimental): BEI intervention that also combines automated text message reminders to dose for insulin; will test Contingent and Non-Contingent BEI
  Interventions: Behavioral: Coin2Dose
- Standard Care Control (No Intervention): Standard care control group; will not receive automated text message reminders to dose for insulin nor BEI for daily BOLUS scores

INTERVENTIONS:
Behavioral: Coin2Dose — Behavioral Economics incentive intervention that also combines automated text message reminders to dose for insulin
  Arms: Coin2Dose

SUMMARY:
Our objective is to test the feasibility, acceptability, and initial efficacy of using behavioral economics incentives (BEI) in a novel, semi-automated intervention to target daily insulin BOLUS scores in adolescents with suboptimal insulin use.

DETAILED DESCRIPTION:
This R01 responds to PAS-20-160 (Small R01s for Clinical Trials Targeting Diseases within the Mission of NIDDK). Our objective is to test the feasibility, acceptability, and initial efficacy of using behavioral economics incentives (BEI) in a novel, semi-automated intervention to target daily insulin BOLUS scores in adolescents with suboptimal insulin use. There is a critical need for efficacious and easy to implement interventions targeting self-management behaviors in adolescents with type 1 diabetes (T1D). This is because national registry data suggest that only between 15-28% of adolescents achieve their glycated hemoglobin (HbA1c) target, thereby placing the majority of them at increased risk for serious acute and long-term complications. BEI interventions are efficacious for promoting health behaviors including frequency of self-monitoring blood glucose (SMBG) in youth. Moreover, there is evidence that BEI can be relatively easy to implement, especially when using Non-Contingent BEI. But with the uptake of integrated insulin pump and continuous glucose monitor (CGM) systems and the new FDA approval enabling youth to dose for insulin based solely on CGM, we believe the long-term value of targeting SMBG alone in BEI interventions is limited and that daily insulin use is the next logical self-management target. Building off of our prior work, the insulin BOLUS score offers a specific, measurable, and valid treatment target for daily insulin use that is also more closely related to HbA1c than SMBG or Total insulin boluses per day. Thus our Aims are: 1) examine the feasibility and acceptability of our semi-automated BEI intervention (called Coin2Dose) that targets daily BOLUS scores in adolescents and 2) examine the preliminary efficacy of Coin2Dose versus a standard care control (SC) group on youth daily BOLUS scores, HbA1c, and glucose time in range (TIR). We also include an exploratory aim to examine the incremental impact of using Contingent versus Non-Contingent BEI within our Coin2Dose intervention on youth's BOLUS scores, HbA1c, and TIR. Coin2Dose will deliver automated text messages to cue adolescents to bolus for insulin, plus BEI for daily BOLUS activity. To enhance the scientific rigor of this R01, we will use the ORBIT Model for behavioral intervention development. Consistent with this model, we will recruit 180 adolescents and a parent to participate in 1- a telehealth focus group (ORBIT Phase 1a: Define; n= 20), 2- a formative pre-test (ORBIT Phase 1b: Refine; n=10), or 3- a pilot randomized clinical trial (ORBIT Phase 2: RCT Pilot; n=150). Our RCT Pilot will randomize teens with suboptimal insulin use (BOLUS score <2.5; 70% of teens based on pilot data) to a SC or 1 of 2 versions of Coin2Dose that only differ based on our use of personalized (Contingent) v. non-personalized (Non-Contingent) BEI. Adolescents will participate in 12-weeks of active treatment, plus a 12-week follow-up period. This small R01 is Significant for its potential to yield: 1- preliminary data supporting our new BEI intervention targeting daily BOLUS scores, which may also improve youth HbA1c, 2- novel data exploring the incremental impact of Contingent v. Non-Contingent BEI, which has implications for Coin2Dose as well as the broader uptake of BEI interventions.

ELIGIBILITY:
Inclusion Criteria:

* adolescents between 11.0-17.0 years old and their parent/guardian;
* adolescents have a physician confirmed diagnosis of type 1 diabetes of at least 6 months duration;
* adolescents use an insulin pump for daily type 1 diabetes self-management;
* adolescents evidence sub-optimal daily BOLUS scores (a mean daily BOLUS score <2.5)

Exclusion Criteria:

* adolescents who do not use an insulin pump; adolescents who have an allergy or sensitivity to the adhesive and/or skin preparation used for CGM;
* adolescents with a comorbid chronic condition (e.g., renal disease);
* adolescents and parents who do not speak English

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nemours Children's Health, Jacksonville, Florida
  - Children's Mercy Kansas City, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Undecided
Undecided. Will not share data that may make it possible to identify individual participants.

REFERENCES:
- [Derived] Patton SR, Fox L, Cushing CC, McDonough R, Clements MA. Cash-Only INcentives to promote insulin DOSE engagement: A protocol paper for the pilot randomized controlled trial of COIN2DOSE. Contemp Clin Trials. 2022 Dec;123:107008. doi: 10.1016/j.cct.2022.107008. Epub 2022 Nov 14. PMID 36396067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited participants from 2023-2024. We included youth between 11-17.99 years old with a physician confirmed type 1 diabetes diagnosis of at least 6 months duration prior to study enrollment. Youth needed to be using an insulin pump or Bluetooth connected insulin pen. Parents were eligible if they consented to participate and had a youth who met our inclusion criteria.
  We used both in-clinic and remote recruitment procedures through a national registry.
Pre-assignment Details: After obtaining parent informed consent and permission and youth assent, we enrolled youth in a brief run-in period so they could practice sharing device data with the study team. Once youth had successfully shared two weeks of data, they moved on to complete the baseline assessment. We randomized youth following completion of the baseline assessment. Eighteen youth did not complete the run-in period and therefore did not continue with the trial.
Groups:
- Standard Care: Adolescents randomized to standard care received a weekly text message reminder to share insulin pump or Bluetooth connected insulin pen data with the research team. Youth received up to $2.00/week * 12 weeks for sharing their data with the research team.
- Coin2Dose: Adolescents randomized to Coin2Dose received weekly automated text message reminders to bolus when eating, a text message reminder to share their data with the study team, and a cash incentive for bolusing insulin at mealtimes and sharing their data. Adolescents received up to $17.50 * 12 weeks. Within this group, adolescents either received a personalized cash incentive for bolusing (Contingent) or a non-personalized cash incentive for bolusing (Non-Contingent). To ensure equality in the total amount of money paid to youth in the Contingent and Non-Contingent arms, we applied a yoked control design.
Period: Overall Study
Arm/Group | Standard Care | Coin2Dose
Started | 53 | 102
Completed | 47 | 92
Not Completed | 6 | 10
Not completed — Lost to Follow-up | 6 | 10

BASELINE CHARACTERISTICS:
Population: Participants who successfully completed the run-in period also needed to complete the baseline assessment before we randomized them. There are no differences between these values and the number of participants assigned to groups in the Participant Flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Coin2Dose | Total
Number analyzed (Participants) | 53 | 102 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] — Self-reported youth age in years
  years | 13.92 (1.96) | 13.77 (2.00) | 13.83 (1.98)
Sex: Female, Male [Count of Participants; unit: Participants] — Self-reported youth sex assigned at birth
  Participants
    Female | 26 | 46 | 72
    Male | 27 | 56 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported youth race
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 1 | 3 | 4
    White | 50 | 95 | 145
    More than one race | 2 | 2 | 4
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported youth ethnicity
  Participants
    Hispanic or Latino | 4 | 6 | 10
    Not Hispanic or Latino | 49 | 96 | 145
    Unknown or Not Reported | 0 | 0 | 0
Baseline daily insulin Bolus score [Mean (Standard Deviation); unit: score on a scale] — Calculated using insulin pump data. Count number of mealtime insulin boluses administered within pre-defined time windows. Daily score can range between 0 (no mealtime boluses) and 3 (bolus administered for 3 meals). Calculate an average of daily scores over 7 days. Possible range: 0-3, higher scores indicate more insulin use.
  score on a scale | 2.03 (0.79) | 1.79 (0.89) | 1.87 (0.86)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Hemoglobin- HbA1c
Description: proxy measure of average glycemic levels
Time Frame: change in week 0 outcome at week 13
Population: Lost to follow between baseline and post-treatment: 3 youth assigned to standard care; 4 youth assigned to Coin2Dose
Measure: Mean (Standard Deviation); unit: Change in A1c (%)
Arm/Group | Standard Care | Coin2Dose
Number analyzed (Participants) | 50 | 98
Change in A1c (%) | -0.14 (0.58) | -0.09 (0.65)

2. Primary Outcome: Change in Daily Insulin Bolus Score
Description: valid, objective measure of insulin use in youth with type 1 diabetes; range 0-3, higher scores reflect greater adherence to mealtime insulin use
Time Frame: change in week 0 outcome at week 13
Population: Lost to follow from baseline to post-treatment: 3 youth assigned to standard care; 4 youth assigned to Coin2Dose. There was also a data attribution issue between June 6 and July 24, 2024 that affected our ability to accurately link youth with their insulin pump data. We do not include BOLUS data from youth impacted by this issue.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Standard Care | Coin2Dose
Number analyzed (Participants) | 45 | 88
score on scale | -0.11 (0.56) | -0.08 (0.66)

3. Secondary Outcome: Change in Glucose Time in Range (70-180 mg/dL)
Description: Change in percent time spent with glucose levels between 70-180mg/dL. Time in Range (TIR) data were unavailable for all participants due to unresolved legal/contractual barriers with external CGM vendors. Efforts to resolve these issues are ongoing, we will update with results if data access becomes possible.
Time Frame: change in week 0 outcome at week 13
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: Baseline until end of follow-up, up to 12 weeks
Description: No differences. Applied the same definitions as provided by clinicaltrials.gov.
Arm/Group | Standard Care | Coin2Dose
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/102
Other Adverse Events (participants affected / at risk) | 0/53 | 0/102

LIMITATIONS AND CAVEATS:
Between June 6 and July 24, 2024, a data attribution issue occurred that affected our ability to accurately link youth participants with their insulin pump data. Data from participants impacted by this issue are not included in the current dataset.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT05280184/Prot_SAP_000.pdf